CLINICAL TRIAL: NCT05535608
Title: The Impact of a Natural Ingredients and App Based Intervention Targeting the Nine Hallmarks of Aging on DNA Methylation
Brief Title: Targeting the Nine Hallmarks of Aging on DNA Methylation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TruDiagnostic (Industry)
Collaborators: SRW (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 10349
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRW Cel system (Experimental): Cel1, Cel2, Cel3
  Patients will take all three supplements once daily. Patients will take 2 capsules of each supplement in the morning with food.
  Interventions: Dietary Supplement: SRW Cel System

INTERVENTIONS:
Dietary Supplement: SRW Cel System — Dietary supplement

SUMMARY:
SRW Laboratories has formulated the Cel System protocol, a group of three formulas designed to interact with each of the 9 Hallmarks of Aging and combined this with an App that supports positive lifestyle changes, with a view that, if we can positively impact each Hallmark, we can support healthy aging.

DETAILED DESCRIPTION:
This study will measure the impact of the Cel System protocol on the biological clocks of the participants, as well as measure established biomarkers associated with the 9 Hallmarks and note any aesthetic changes you may experience to establish evidence of the effect of the Cel System Protocol over time.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of any ethnicity
* 55 years and older
* Female subjects must be post-menopausal
* Participant must be able to comply with treatment plan and laboratory tests
* Participant must be able to read, write, and speak English fluently
* Participant must have a smartphone and be able to download and use the App
* Participant must have an established primary care provider
* Participant must be willing and able to consume study supplements throughout the duration of study period

Exclusion Criteria:

* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Known immune system issues or immunodeficiency disease
* History of viral illness which could be reactivated by immune downregulation
* Presence of clinically significant acute or unstable cardiovascular and cerebrovascular (stroke) disease
* Diagnosis of a transient ischemic attack in the 6 months prior to screening
* Participants infected with hepatitis C or HIV
* Presence of active infection in previous 4 weeks
* Any other illness, psychiatric disorder, alcohol or chemical dependence that in the opinion of the Clinical Investigator would render a participant unsuitable to participate in the study
* Unable or unwilling to provide required blood sample for testing
* Current or previous use of known prescription immunomodulating products (e.g. glucocorticoids, TNF-alpha inhibitors) in the month prior to the start of the trial.
* A known history of blood dyscrasias including coagulopathy
* Any person deemed by the Investigator as having a low likelihood of complying with study protocol (e.g. evidence of history of non-compliance, history of poor follow-up, multiple or complex scheduling conflicts).
* Planned surgical procedure during study period
* Participants who are actively engaged in a weight loss program or have started any new medications during the duration of the trial that can potentially interfere with the study, as deemed appropriate by Principal Investigator.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Biological age | Change in epigenetic age from baseline to 12 months
  The primary outcome measure for the study is biological age, measured by DNA methylation, using blood and saliva samples collected from patients.

SECONDARY OUTCOMES:
Inflammatory marker IL-6 | Change in inflammatory marker from baseline to 12 months
  (IL-6 will also be assessed at 3, 6, and 12 months.
C-reactive protein | Change in inflammatory marker from baseline to 12 months
  C-reactive protein will also be assessed at 3, 6, and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Wellness Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blagosklonny MV. Cell senescence, rapamycin and hyperfunction theory of aging. Cell Cycle. 2022 Jul;21(14):1456-1467. doi: 10.1080/15384101.2022.2054636. Epub 2022 Mar 31. PMID 35358003
- [Background] Bungau S, Vesa CM, Abid A, Behl T, Tit DM, Purza AL, Pasca B, Todan LM, Endres L. Withaferin A-A Promising Phytochemical Compound with Multiple Results in Dermatological Diseases. Molecules. 2021 Apr 21;26(9):2407. doi: 10.3390/molecules26092407. PMID 33919088
- [Background] Gonzales MM, Garbarino VR, Marques Zilli E, Petersen RC, Kirkland JL, Tchkonia T, Musi N, Seshadri S, Craft S, Orr ME. Senolytic Therapy to Modulate the Progression of Alzheimer's Disease (SToMP-AD): A Pilot Clinical Trial. J Prev Alzheimers Dis. 2022;9(1):22-29. doi: 10.14283/jpad.2021.62. PMID 35098970
- [Background] Hong W, Mo F, Zhang Z, Huang M, Wei X. Nicotinamide Mononucleotide: A Promising Molecule for Therapy of Diverse Diseases by Targeting NAD+ Metabolism. Front Cell Dev Biol. 2020 Apr 28;8:246. doi: 10.3389/fcell.2020.00246. eCollection 2020. PMID 32411700
- [Background] Hassan FU, Rehman MS, Khan MS, Ali MA, Javed A, Nawaz A, Yang C. Curcumin as an Alternative Epigenetic Modulator: Mechanism of Action and Potential Effects. Front Genet. 2019 Jun 4;10:514. doi: 10.3389/fgene.2019.00514. eCollection 2019. PMID 31214247